CLINICAL TRIAL: NCT07072962
Title: TeleExergame: Remotely-supervised Exercise Platform for Improving Cognition and Motor Function Using Telemedicine - Phase I
Brief Title: Self-Administered Interactive Exercise Program (Tele-Exergame)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH); BioSensics (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-44913 - Phase I; R44AG067909 (NIH)
Record Dates: First submitted 2025-06-25; First posted 2025-07-18 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment (MCI); Mild Alzheimer Disease; Memory Deficits
Keywords: exercise; interactive exercise; exergame; tele-rehabilitation; home-based exercise; telemedicine; wearables; cognitive impairment; dementia; balance; telehealth; Alzheimer's disease; gamification
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Motor Activity; Dementia

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention: a self-administered home exercise program delivered via an interactive tablet-based system (Tele-Exergame) designed to provide supportive care for individuals with mild cognitive impairment or early dementia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TeleExergame (Experimental): Participants assigned to the Tele-Exergame arm will engage in a tablet-based, home-delivered exercise program focused on foot and ankle mobility, designed specifically for older adults with cognitive impairment or mild dementia. The intervention aims to enhance balance, mobility, and cognitive engagement through structured and gamified motor exercises.
  Each session includes a sequence of guided exercises such as ankle dorsiflexion and plantarflexion and seated marching, with an emphasis on safe, repetitive movement. Sessions are conducted two times per week, lasting approximately 20-30 minutes each, over a period of 6 weeks.
  Instructional cues are provided via synchronized audio, images, and text on a user-friendly tablet interface. A motion sensor worn on the foot tracks movement in real time, delivering instant feedback on range of motion and task completion. Exercise performance and adherence data are securely transmitted to a cloud-based server for remote remote monitoring.
  Interventions: Device: home-based self-administered interactive exercise

INTERVENTIONS:
Device: home-based self-administered interactive exercise — The Tele-Exergame system delivers a structured foot and ankle exercise program tailored for individuals with cognitive impairment or mild dementia to support balance and cognitive function. Exercises such as leg raising and foot flexion are guided through audio, visual, and text prompts on a tablet. A foot-mounted motion sensor provides real-time feedback to ensure proper range of motion, while exercise data are securely streamed to the cloud for remote monitoring of adherence. The system also includes a telemedicine interface to enable remote support and education when needed.
  Other Names: Teleexergame

SUMMARY:
This longitudinal Phase I feasibility trial combines care-as-usual with a 6-week, single-arm exercise intervention using Tele-Exergame, an interactive, self-administered home-based exercise program aimed at improving cognitive-motor function in individuals with mild cognitive impairment (MCI) and dementia. Fifteen participants will complete two 30-minute sessions per week via the Tele-Exergame platform. Outcomes will be assessed at baseline and post-intervention, with the primary outcome being change in cognition. Secondary outcomes include acceptability, dropout rate, and changes in anxiety.

DETAILED DESCRIPTION:
At the beginning of the 6-week in-home exergaming intervention using the proposed Tele-Exergame system, participants will complete baseline assessments to evaluate system acceptance, cognitive function, and anxiety levels. Acceptance will be measured using the Technology Acceptance Model (TAM) questionnaire-a validated, intention-based Likert scale tool assessing user satisfaction with technology-comprising 11 items (two on ease of use, seven on perceived benefit, and two on attitudes toward use). Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), and anxiety levels will be evaluated using the Beck Anxiety Inventory (BAI). Participants will be instructed to perform leg-raising or foot-flexion exercises, guided by the Tele-Exergame platform, for approximately 30 minutes twice per week over six consecutive weeks. Motion sensors (a motion sensor, which is part of of the Tele-Exergame system) will be worn on the upper leg for leg-raising exercises and on the foot for foot-flexion exercises. At the end of the 6-week intervention, participants will complete post-assessments for acceptance, cognition, and anxiety using the same measures.

ELIGIBILITY:
Inclusion Criteria:

* Are 50 years of age or older,
* Have a clinical diagnosis of mild cognitive impairment (MCI) or dementia, or a MoCA score of 25 or below indicating cognitive decline,
* Are able to walk at least 20 meters, with or without assistance,
* Live independently in a residential setting with access to a caregiver or informant, and
* Are willing and able to provide informed consent

Exclusion Criteria:

* Have severe mobility limitations or conditions that prevent safe participation in a weight-bearing exercise program (e.g., double amputation, active foot ulcers, or significant pain in the back or lower extremities),
* Have severe cognitive impairment that may limit their ability to interact with tablet.
* Have a recent neurological condition (less than 6 months) known to affect cognition (e.g., stroke, Parkinson's disease, traumatic brain injury)
* Have a significant psychiatric disorder, current substance abuse, or any medical condition that would interfere with study participation, or
* Have major hearing or vision impairment limit their ability to interact with the device

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This study was submitted as part of an NIH SBIR project with a subaward from BioSensics LLC. Individual-level data will be shared with permission from BioSensics LLC based on the contract agreement. However, aggregated results for all participants will be published and reported.

REFERENCES:
- [Result] Park C, Mishra RK, York MK, Enriquez A, Lindsay A, Barchard G, Vaziri A, Najafi B. Tele-Medicine Based and Self-Administered Interactive Exercise Program (Tele-Exergame) to Improve Cognition in Older Adults with Mild Cognitive Impairment or Dementia: A Feasibility, Acceptability, and Proof-of-Concept Study. Int J Environ Res Public Health. 2022 Dec 6;19(23):16361. doi: 10.3390/ijerph192316361. PMID 36498431

RESULTS

PARTICIPANT FLOW:
Groups:
- TeleExergame: Participants in the Tele-Exergame arm will use a home-based, tablet-guided exercise program, called TeleExergame, designed to improve foot and ankle mobility, balance, and cognitive function in older adults with cognitive impairment or mild dementia. The 6-week program consists of two 20-30 minute sessions per week, featuring safe, repetitive exercises such as foot flexion, ankle dorsiflexion, and seated marching. Instructions are provided through synchronized audio, visual, and text prompts. A foot-worn motion sensor tracks movements in real time, offering immediate feedback and securely transmitting adherence and performance data to a cloud server for remote monitoring. The system also supports telemedicine-based coaching and education when needed.
Period: Overall Study
Arm/Group | TeleExergame
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- TeleExergame: Participants used a home-based, tablet-guided exercise program, called TeleExergame, designed to improve foot and ankle mobility, balance, and cognitive function in older adults with cognitive impairment or mild dementia. The 6-week program consists of two 20-30 minute sessions per week, featuring safe, repetitive exercises such as foot flexion, ankle dorsiflexion, and seated marching. Instructions are provided through synchronized audio, visual, and text prompts. A foot-worn motion sensor tracks movements in real time, offering immediate feedback and securely transmitting adherence and performance data to a cloud server for remote monitoring. The system also supports telemedicine-based coaching and education when needed.
Arm/Group | TeleExergame
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Cognitive Function at 6 Weeks Compared to Baseline
Description: Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a validated 30-point screening tool designed to detect mild cognitive impairment and early dementia. The MoCA evaluates multiple cognitive domains, including memory, attention, language, visuospatial abilities, executive function, and orientation. Scores range from 0 to 30, with higher scores indicating better cognitive performance. The MoCA will be administered at baseline and at 6 weeks. The outcome will be reported as the percentage change in total MoCA score from baseline to 6 weeks, calculated as:
  [(Week 6 Score - Baseline Score) / Baseline Score] × 100. A positive percentage indicates improved cognitive performance.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- TeleExergame: Participants iused a home-based, tablet-guided exercise program, called TeleExergame, designed to improve foot and ankle mobility, balance, and cognitive function in older adults with cognitive impairment or mild dementia. The 6-week program consists of two 20-30 minute sessions per week, featuring safe, repetitive exercises such as foot flexion, ankle dorsiflexion, and seated marching. Instructions are provided through synchronized audio, visual, and text prompts. A foot-worn motion sensor tracks movements in real time, offering immediate feedback and securely transmitting adherence and performance data to a cloud server for remote monitoring. The system also supports telemedicine-based coaching and education when needed.
Arm/Group | TeleExergame
Number analyzed (Participants) | 12
percentage change | 9.7 (10.8)

2. Secondary Outcome: Acceptability
Description: To evaluate participant acceptance of the Tele-Exergame system, the Technology Acceptance Model (TAM) questionnaire was administered. TAM is an intention-based framework widely used to assess user satisfaction and acceptance of new technologies. The questionnaire included 31 items: 15 assessed perceived ease of use, 11 evaluated perceived benefits, and 5 measured attitudes toward use. Responses were rated on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree), resulting in a total score range of 0 to 124. A score of 93 or higher was considered indicative of an acceptable level of program acceptance.
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TeleExergame
Number analyzed (Participants) | 12
score on a scale | 93.3 (17.4)

3. Secondary Outcome: Percentage Change in Anxiety Levels at 6 Weeks Compared to Baseline
Description: Anxiety will be assessed using the Beck Anxiety Inventory (BAI), a 21-item self-report questionnaire that measures the severity of anxiety symptoms. Each item is scored on a scale from 0 (not at all) to 3 (severely), resulting in a total score ranging from 0 to 63, with higher scores indicating greater anxiety. The BAI will be administered at baseline and at 6 weeks. The outcome will be reported as the percentage change in total BAI score from baseline to 6 weeks, calculated as:
  [(Week 6 Score - Baseline Score) / Baseline Score] × 100. A negative percentage indicates a reduction in anxiety symptoms
Time Frame: baseline and week 6
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TeleExergame
Number analyzed (Participants) | 12
percentage change | -52.4 (40.3)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The following adverse events were monitored: muscle strain, joint pain, tendonitis, cramps, dizziness, headache, palpitations, chest discomfort, shortness of breath, falls, sprains, nausea, fatigue, weakness, excessive sweating, and exercise intolerance. Serious events included dementia progression, hospitalization, accidents preventing exercise, and death.
Arm/Group | TeleExergame
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This is an NIH SBIR grant with BioSensics LLC as the prime awardee. A subaward contract agreement between BioSensics LLC and Baylor College of Medicine is in place, which may restrict the sharing of certain results deemed confidential.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT07072962/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT07072962/ICF_001.pdf